CLINICAL TRIAL: NCT04410874
Title: MVA-BN Imvamune Smallpox Vaccine Virus for Treatment of Basal Cell Carcinoma, Squamous Cell Carcinomas
Brief Title: Imvamune Vaccine for the Treatment of Non-melanoma Skin Cancer
Acronym: MUSIC-01
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inability to recruit patients/lack of funding
Sponsor: Ivan Litvinov (Other)
Responsible Party: Sponsor-Investigator, Ivan Litvinov, Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-4599
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Non-melanoma Skin Cancer; Basal Cell Carcinoma; Squamous Cell Carcinoma
Keywords: Skin Cancer; Immunotherapy
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Skin Neoplasms | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imvamune (Experimental): Imvamune vaccine to be administered intratumorally at one of three doses on Days 0 and 4 of the study
  Interventions: Biological: Imvamune

INTERVENTIONS:
Biological: Imvamune — Imvamune vaccine to be administered (via injection) intratumorally at one of three doses (1x10^7, 1x10^8, or 4x10^8 PFU) twice, 4 days apart (first injection on Day 0 of the study and second injection on Day 4)
  Other Names: MVA-BN Smallpox vaccine; Modified Vaccinia Ankara Smallpox Vaccine

SUMMARY:
This study examines the safety and efficacy of using the Imvamune smallpox vaccine in the treatment of non-melanoma skin cancers (basal cell carcinoma and squamous cell carcinoma).

DETAILED DESCRIPTION:
One of the main ways cancer is able to develop is by hiding or evading our immune system which usually detects and kills potential tumor cells. Once cancer has developed the ability to evade the immune system it can continue to grow and become a tumor. One potential strategy currently being researched, called immunotherapy, uses viruses to stimulate an immune response which attacks the tumor.

Imvamune is a live, non-replicating virus used in Canada to vaccinate adults and children against smallpox. It is safe to use in immunosuppressed patients because the virus is unable to replicate and spread past the first infected cell. This makes the Imvamune vaccine a viable candidate for immunotherapy in immunosuppressed patients who are at a much higher (up to 60x) risk of developing non-melanoma skin cancers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed, BCC and/or SCC tumors located on the chest, back, thigh, or arm/forearm.
* Presence of clinically documented disease. Skin tumor should measure at least 10 mm in size and should be no larger than 5 cm in any axes. There should be no clinical suspicion of metastasis (i.e. no lymphadenopaties and no systemic symptoms).
* Age > 18 years.
* Subjects must have a documented ECOG performance status of 0 or 1.
* Subjects could be treatment naive or could have had previous surgery or radiation
* Subjects may have had prior radiation therapy. A minimum of 28 days (4 weeks) must have elapsed between the last dose of radiation and date of registration (14 days for a single palliative fraction of radiation to a non-target lesion). Subjects must have recovered from any acute toxic effects from radiation prior to registration (unless grade 1, irreversible and considered not clinically significant).
* Previous surgery is permitted. A minimum of 28 days (4 weeks) must have elapsed between any major surgery and date of registration (7 days for minor surgery), provided that wound healing has occurred
* Each subject must sign a consent form prior to registration/at registration and prior to tests which are study specific.
* Subjects must be accessible for treatment and follow-up. Subjects registered on this trial must be treated and followed at the McGill University Health Centre (MUHC) or McGill Affiliated/other participating hospitals
* Laboratory requirements (must be done within 7 days prior to registration or at time of registration) as follows:
* White blood cell count ≥3.0x10^9/L
* absolute neutrophils ≥1.5x10^9/L
* hemoglobin ≥100g/L
* platelets ≥75x10^9/L
* INR ≤1.2
* bilirubin ≤1.5x upper normal limit
* AST and ALT ≤3.0x upper normal limit
* serum creatinine ≤1.5x upper normal limit (or creatinine clearance of ≥60mL/min)

Exclusion Criteria:

* Cancers located on cosmetically/functionally important areas (i.e. face, neck, genitalia, hands, feet, and lower legs).
* Tumor larger than 5 cm in size (any axes).
* Metastatic disease (or suspicion of metastasis).
* Tumors arising as part of a genetic syndrome (i.e., Bazex-Dupré-Christol, Basal Cell Nevus Syndrome, Rombo syndromes for BCC or Xeroderma Pigmentosa, Ferguson Smith, Grzybowski, Muir-Tore syndromes for SCC).
* Immunosuppressed individuals (e.g. organ transplant recipients, patient with inherited immunodeficiencies, HIV+ individuals or individuals receiving immunosuppressive medications for other reasons).
* Individuals that are not able or willing to sign an informed consent.
* Subjects with history of other active or current malignancies requiring active treatment.
* Patients undergoing concurrent treatments with other anti-cancer therapy or other investigational agents.
* Subjects with prior treatment with Imvamune
* Subjects with serious illness or medical condition that would not permit management
* Subjects with uncontrolled pre-existing cardiovascular conditions and/or symptomatic cardiac dysfunction.
* Pregnant or lactating women. Men or women of childbearing potential who do not agree to use adequate contraception while on trial and 6 weeks following the trial.
* Subjects using anti-viral medications, steroids, immunosuppressive agents, or immunization (including the flu shot) within 14 days prior to registration. Patients who are at high risk of influenza infection (65 years and older, people of any age with certain chronic medical conditions (such as asthma, diabetes, or heart disease), pregnant women and children younger than 5 years), and who have not received an influenza vaccination during the flu season (i.e., October to May).
* Subjects with a condition that could have resulted in splenic dysfunction (e.g. splenectomy, sickle cell anemia, radiation to the spleen ≥ 20Gy, congenital asplenism).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 25 days
  The MTD will be defined as the dose at which 2 or more patients experience a grade 3 or 4 adverse event (as defined by NCI Common Terminology Criteria for Adverse Events version 5.0) that is at least "probably related" to the study drug (ex: dose limiting toxicity).
Objective Tumor Response Rate (ORR) | 25 days
  Clinical and histological evaluation of the tumor to assess the development of immunity against BCC and/or SCC tumors or their protein markers.

SECONDARY OUTCOMES:
Viral load in NMSC tumours | 25 days
  Ability to detect viral infection in the tumor.
Number of T cells/concentration of antigen specific antibodies | 25 days
  Ability to elicit increased immunological T/NKT cell mediated response, and antibody response against the tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan V Litvinov, M.D., Ph.D, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No